CLINICAL TRIAL: NCT01037582
Title: Investigation on Safety, Tolerability and Bioavailability of Oral NN9924 in Healthy Male Subjects
Brief Title: A Two Part Trial Investigating the Safety of NN9924 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-3691; 2009-012366-31 (EudraCT Number); U1111-1112-7564 (Other: WHO)
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial part 1 (Experimental)
  Interventions: Drug: NN9924 (oral); Drug: placebo
- Trial part 2 (Experimental)
  Interventions: Drug: NN9924 (oral); Drug: placebo; Drug: NN9924 (s.c.); Drug: NN9924 (i.v.)

INTERVENTIONS:
Drug: NN9924 (oral) — Subjects will be randomized to receive a single dose of NN9924, at escalating dose levels. Progression to next dose will be based on safety evaluation.
  Arms: Trial part 1
Drug: placebo — Subjects will receive a single dose of placebo as a comparator to NN9924, at all dose levels.
  Arms: Trial part 1
Drug: NN9924 (oral) — Subjects will be randomized to receive a single dose of NN9924 in one of three different concentrations. The dose will be selected based on the results of part 1.
  Arms: Trial part 2
Drug: placebo — Subjects will be randomized to receive a single dose of placebo.
  Arms: Trial part 2
Drug: NN9924 (s.c.) — As an active comparator, one standard dose will be given s.c. (under the skin) at one study visit
  Arms: Trial part 2
Drug: NN9924 (i.v.) — As an active comparator, one standard dose will be given i.v. (into the vein) at one study visit.
  Arms: Trial part 2

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the safety, tolerability and bioavailability (exploring absorption of drug in body) of NN9924 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with good general health as judged by the Investigator
* Body weight of 65.0-95.0 kg (both inclusive)
* Body Mass Index (BMI) of 18.5-27.5 kg/m^2 (both inclusive)

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Acute infection or inflammation or other illness that may confound the results of the trial or pose a risk to the subject by administering the trial product, as judged by the Investigator
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea) or malabsorptive states (celiac disease, lactose intolerance or chronic pancreatitits), as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2009-12-17 (Actual); Primary Completion 2010-05-07 (Actual); Study Completion 2010-05-07 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events (AEs) recorded | from dosing to Day 22

SECONDARY OUTCOMES:
The uptake in blood of oral NN9924 compared to i.v. and s.c. administration of the same compound | from 0 to 504 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Harrow, United Kingdom

REFERENCES:
- [Derived] Granhall C, Donsmark M, Blicher TM, Golor G, Sondergaard FL, Thomsen M, Baekdal TA. Safety and Pharmacokinetics of Single and Multiple Ascending Doses of the Novel Oral Human GLP-1 Analogue, Oral Semaglutide, in Healthy Subjects and Subjects with Type 2 Diabetes. Clin Pharmacokinet. 2019 Jun;58(6):781-791. doi: 10.1007/s40262-018-0728-4. PMID 30565096
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com